CLINICAL TRIAL: NCT01145274
Title: A Pilot Study for PK/PD Parameter of Allopurinol and Its Metabolite-oxypurinol After Once-daily Allopurinol in Chronic Kidney Disease Patient
Brief Title: A Pilot Study for Pharmacokinetic/Pharmacodynamic (PK/PD) Parameter of Allopurinol and Its Metabolite-oxypurinol After Once-daily Allopurinol in Chronic Kidney Disease Patient
Acronym: Allopurinol
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Suhnggwon Kim, Seoul National University Hospital
Other Study IDs: Allopurinol_2010_1
Record Dates: First submitted 2010-06-15; First posted 2010-06-16 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2011-08

CONDITIONS: Chronic Kidney Disease
Keywords: allopurinol; chronic kidney diseae
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
To know the blood level of allopurinol in chronic kidney disease (CKD) patient.

DETAILED DESCRIPTION:
After the result of this pilot study, we can prescribe the optimal dose of allopurinol in CKD patient.

ELIGIBILITY:
Inclusion Criteria:

* from 18yrs to 80yrs , man and women
* the patient who are taking allopurinol
* On screening, the patient shows that the level of protein/creatinine ratio is over 3.0
* On screening, the patient shows that MDRD GFR >= 30 ml/min and <= 60 ml/min
* the patient sign on the concent form

Exclusion Criteria:

* the patient have experience to take medication that have an effect on renal function
* the patient have experience to take cyclosporin within 3month
* At least, the average level of two separate blood pressure ( 2min interval ) shows that SBP <= 100 mmHg or >=160 mmHg and DBP <=60 mmHg >=100 mmHg, or Heart rate < 40 beats/min or > 90 beats/min
* uncontrolled hypertension
* pregnancy or anticipate pregnancy with 6 month
* hypersensitivity to allopurinol
* acute hepatitis or the level of AST or ALT is over 2times of normal range or the level of bilirubin is over 2.0 mg/dL
* serum albumin < 3.5 mg/dL or > 5mg/dL
* urinary retension, prostatic hyperplasia
* the patient show gout attack on taking allopurinol
* the patient who have gastro-intestinal disease ( ex, crohn's disease, acute or chronic pancreatitis, ulcer )or who have the surgical history of gastrointestine.
* the patient who should take azathioprine, mercaptopurine, cyclophosphamide, Losartan, benzbromarone,fenofibrate,furosemide ,probenecid
* the patient who had taken part in the other study within 3months
* the patient who had gotten blood transfusion
* pregnant, breast feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: chronic kidney disease ( estimated GFR 30-60 ml/min )
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2010-06; Primary Completion 2013-02 (Estimated); Study Completion 2013-02 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea